CLINICAL TRIAL: NCT01254006
Title: Retinal Nerve Fibres Layers Thickness Study in Glaucomatous Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Roma La Sapienza (Other)
Collaborators: vingolo enzo maria (Unknown); domanico daniela (Unknown); salvatore serena (Unknown)
Other Study IDs: GLA0110
Record Dates: First submitted 2010-11-29; First posted 2010-12-06 (Estimated); Last update posted 2010-12-06 (Estimated); Status verified 2009-08

CONDITIONS: Glaucoma
MeSH Terms: conditions — Glaucoma | interventions — Colforsin; Rutin

INTERVENTIONS:
Drug: forskolin, rutin and vitamins B1 and B2

SUMMARY:
In this study the investigators are going to study the retinal nerve fibers layers (RNFL) modification of two groups of patients, one taking no drugs, the other taking forskolin, rutin and vitamins B1 and B2.

ELIGIBILITY:
Inclusion Criteria:

* Age (30-80 years);
* Baseline Intraocular pressure (IOP) (20-32 mmHg): average untreated Intra Ocular Pressure (IOP) for both eyes as determined from 2 to 4 visits within a 6-months period;
* Central Corneal Thickness (CCT) (475-650 µm): average of 3 different measurements from both eyes during the same visit;
* Pattern standard deviation (PSD) (0,50-3,00 dB) average of both eyes as stated on the most recent visual field index report
* Vertical Cup/Disk ratio (0,00-0,80): average of both eyes
* All these data were entered into a calculator specially designed for STAR (Scoring Tool for assessing risk) II parameter. The patients were divided into low-, moderate- and high risk groups according to the result given by the calculator.

Exclusion Criteria:

-other ocular pathologies than glaucoma

Ages: 30 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult

PRIMARY OUTCOMES:
retinal nerve fibres layer thickness

SECONDARY OUTCOMES:
global risk threshold for glaucoma progression

CONTACTS AND LOCATIONS:
Locations (1):
- Univerisity La Sapienza, Latina, Italy